CLINICAL TRIAL: NCT01639157
Title: Human Laboratory Study of the Impact of Buspirone Maintenance on the Reinforcing, Subjective and Performance Effects of Cocaine
Brief Title: Impact of Buspirone Maintenance on the Reinforcing Effects of Cocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: R21DA034095-01 (NIH)
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Cocaine Use Disorders
MeSH Terms: interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buspirone (Experimental): Subjects will be maintained on 30 mg buspirone daily.
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Subjects will be maintained on placebo (i.e., 0 mg buspirone daily).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Subjects will be maintained on oral buspirone (10 mg administered 3 times daily) for 6 days each during the study in random order.
  Arms: Buspirone
Drug: Placebo — Subjects will be maintained on oral placebo (0 mg administered 3 times daily) for 6 days each during the study in random order.
  Arms: Placebo

SUMMARY:
Cocaine use disorders are an unrelenting public health concern. Intensive research efforts have yielded behavioral interventions that reduce cocaine use, however, these interventions are not universally effective and treatment effects diminish over time. Development of a pharmacotherapy that enhances the efficacy of these interventions is a priority for the National Institute on Drug Abuse. This study proposes to determine the impact of buspirone maintenance on self-administration of cocaine and alternative reinforcers. These preliminary data will be used to support further research developing buspirone as a pharmacotherapy for cocaine use disorders. We hypothesize that buspirone will attenuate the reinforcing effects of cocaine and increase the reinforcing effects of alternative reinforcers.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine or buspirone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

REFERENCES:
- [Background] Stoops WW, Lile JA, Glaser PE, Hays LR, Rush CR. Intranasal cocaine functions as reinforcer on a progressive ratio schedule in humans. Eur J Pharmacol. 2010 Oct 10;644(1-3):101-5. doi: 10.1016/j.ejphar.2010.06.055. Epub 2010 Jul 16. PMID 20638380

RESULTS

PARTICIPANT FLOW:
Groups:
- Buspirone Then Placebo: Subjects were maintained on 30 mg buspirone daily for 6 days, then they were crossed over to placebo daily for 6 days.
- Placebo Then Buspirone: Subjects were maintained on placebo daily for 6 days, then they were crossed over to 30 mg buspirone daily for 6 days.
Period: Overall Study
Arm/Group | Buspirone Then Placebo | Placebo Then Buspirone
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Subjects were maintained on oral buspirone (10 mg administered 3 times daily) or placebo for 6 days each during the study in random order.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 39.4 [26 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Times Cocaine Was Selected in the Presence of a Monetary Reward Alternative
Description: The reinforcing effects of cocaine were determined using a modified progressive ratio procedure (Stoops et al., 2010) in which subjects made 6 choices between available each available cocaine dose and money (US$0.25). Reinforcing effects are measured for each cocaine dose during both buspirone and placebo maintenance.
Time Frame: One test per cocaine dose level per intervention for each participant over his/her 2 week inpatient admission
Measure: Mean (Standard Error); unit: Number of Cocaine Choices
Groups:
- Buspirone: Subjects were maintained on 30 mg buspirone daily for 6 days.
- Placebo: Subjects were maintained on placebo daily for 6 days.
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
Number of Cocaine Choices
  0 mg Cocaine | 1.00 (0.707) | 1.22 (0.813)
  15 mg Cocaine | 5.56 (0.338) | 5.33 (0.441)
  45 mg Cocaine | 5 (.289) | 4.89 (.455)

2. Secondary Outcome: Peak Score on Sedative Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Sedative Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "sedative" items was summed to yield the Sedative Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: Subjects completed this measure at 15 minute intervals for 45 minutes after sampling each cocaine dose under both buspirone and placebo maintenance conditions.
Measure: Mean (Standard Error); unit: arbitrary units on a Likert-type scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitrary units on a Likert-type scale
  0 mg Cocaine | 2.9 (1.3) | 3.6 (1.6)
  15 mg Cocaine | 4.4 (1.7) | 4.8 (1.8)
  45 mg Cocaine | 5.6 (1.8) | 3.1 (1.1)

3. Secondary Outcome: Peak Systolic Blood Pressure
Description: Systolic blood pressure was measured with an automated monitor. Higher values represent greater systolic pressure. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: This measure was completed at 15 minute intervals for 45 minutes after sampling each cocaine dose under both buspirone and placebo maintenance conditions.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
mmHg
  0 mg Cocaine | 120.8 (3.3) | 120.6 (3.2)
  15 mg Cocaine | 128.7 (1.3) | 127.0 (3.4)
  45 mg Cocaine | 127.1 (2.9) | 131.8 (3.0)

4. Secondary Outcome: Peak Score on Stimulant Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Stimulant Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "sedative" items was summed to yield the Stimulant Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitrary units on a Likert-type scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitrary units on a Likert-type scale
  0 mg Cocaine | 5 (1.7) | 4.4 (1.1)
  15 mg Cocaine | 9.8 (1.7) | 9 (1.5)
  45 mg Cocaine | 11.4 (2.1) | 11.3 (2.0)

5. Secondary Outcome: Peak Ratings of "Active, Alert, Energetic" on the Visual Analog Scale
Description: Subjects rated their feelings of "Active, Alert, Energetic" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.8 (3.0) | 3.7 (2.9)
  15 mg Cocaine | 20.1 (6.0) | 17.4 (5.4)
  45 mg Cocaine | 24.7 (7.7) | 33.3 (8.3)

6. Secondary Outcome: Peak Ratings of "Any Effect" on the Visual Analog Scale
Description: Subjects rated their feelings of "Any Effect" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 6.2 (4.8) | 6.1 (3.7)
  15 mg Cocaine | 23.0 (4.7) | 17.3 (5.2)
  45 mg Cocaine | 26 (6.5) | 33.4 (8.0)

7. Secondary Outcome: Peak Ratings of "Bad Effects" on the Visual Analog Scale
Description: Subjects rated their feelings of "Bad Effects" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 4.3 (3.5) | 5.9 (3.8)
  15 mg Cocaine | 6.7 (3.0) | 7.7 (2.9)
  45 mg Cocaine | 12.2 (4.8) | 9.1 (4.4)

8. Secondary Outcome: Peak Ratings of "Euphoric" on the Visual Analog Scale
Description: Subjects rated their feelings of "Euphoric" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 5.6 (4.7) | 5.9 (4.9)
  15 mg Cocaine | 15.8 (8.2) | 13.1 (7.4)
  45 mg Cocaine | 16.4 (9.3) | 14.1 (6.9)

9. Secondary Outcome: Peak Ratings of "Good Effects" on the Visual Analog Scale
Description: Subjects rated their feelings of "Good Effects" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 4.8 (3.9) | 3.3 (2.6)
  15 mg Cocaine | 21.3 (4.9) | 15.7 (5.0)
  45 mg Cocaine | 21.2 (6.1) | 32.3 (6.8)

10. Secondary Outcome: Peak Ratings of "High" on the Visual Analog Scale
Description: Subjects rated their feelings of "High" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 5.1 (4.4) | 3.9 (3.4)
  15 mg Cocaine | 17.9 (5.2) | 12.7 (5.0)
  45 mg Cocaine | 21.4 (7.0) | 27.2 (6.0)

11. Secondary Outcome: Peak Ratings of "Irregular/Racing Heartbeat" on the Visual Analog Scale
Description: Subjects rated their feelings of "Irregular/Racing Heartbeat" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.9 (3.3) | 2.3 (1.3)
  15 mg Cocaine | 11.1 (6.3) | 9.1 (6.0)
  45 mg Cocaine | 20.1 (8.4) | 14.3 (4.8)

12. Secondary Outcome: Peak Ratings of "Like Drug" on the Visual Analog Scale
Description: Subjects rated their feelings of "Like Drug" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.6 (2.5) | 2.1 (1.5)
  15 mg Cocaine | 23.9 (6.0) | 18.3 (6.4)
  45 mg Cocaine | 30.3 (8.4) | 36.1 (7.8)

13. Secondary Outcome: Peak Ratings of "Nauseated, Queasy, Sick to Stomach" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nauseated, Queasy, Sick to Stomach" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.8 (3.1) | 1.6 (1.1)
  15 mg Cocaine | 8.8 (5.7) | 10.6 (5.7)
  45 mg Cocaine | 13.4 (6.3) | 11.1 (5.4)

14. Secondary Outcome: Peak Ratings of "Nervous, Anxious" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nervous, Anxious" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.6 (3.0) | 2 (1.4)
  15 mg Cocaine | 13.1 (5.8) | 10.2 (4.6)
  45 mg Cocaine | 17.2 (7.4) | 12.6 (5.2)

15. Secondary Outcome: Peak Ratings of "Willing to Pay For" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Pay For" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.6 (2.7) | 3.1 (2.4)
  15 mg Cocaine | 18.6 (5.4) | 13.9 (4.5)
  45 mg Cocaine | 31.9 (10.9) | 31.3 (8.8)

16. Secondary Outcome: Peak Ratings of "Performance Impaired" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Impaired" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 2.6 (2.1) | 4.3 (2.5)
  15 mg Cocaine | 8.8 (5.2) | 6.3 (3.3)
  45 mg Cocaine | 12.6 (6.8) | 18.2 (8.4)

17. Secondary Outcome: Peak Ratings of "Performance Improved" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Improved" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 2.7 (1.9) | 1.9 (1.3)
  15 mg Cocaine | 8.9 (5.6) | 5.2 (2.8)
  45 mg Cocaine | 4.7 (3.1) | 4.8 (2.7)

18. Secondary Outcome: Peak Ratings of "Restless" on the Visual Analog Scale
Description: Subjects rated their feelings of "Restless" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 4.1 (3.6) | 1.9 (1.2)
  15 mg Cocaine | 10.0 (6.3) | 10.2 (5.0)
  45 mg Cocaine | 13.0 (6.4) | 9.4 (4.4)

19. Secondary Outcome: Peak Ratings of "Rush" on the Visual Analog Scale
Description: Subjects rated their feelings of "Rush" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.6 (2.8) | 1.9 (1.3)
  15 mg Cocaine | 18.4 (5.1) | 12.4 (4.1)
  45 mg Cocaine | 20.1 (5.8) | 23.3 (6.2)

20. Secondary Outcome: Peak Ratings of "Shaky, Jittery" on the Visual Analog Scale
Description: Subjects rated their feelings of "Shaky, Jittery" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 4.8 (4.1) | 2.1 (1.5)
  15 mg Cocaine | 15.1 (6.0) | 11.4 (5.2)
  45 mg Cocaine | 18.9 (8.2) | 17.7 (5.3)

21. Secondary Outcome: Peak Ratings of "Sluggish, Fatigued, Lazy" on the Visual Analog Scale
Description: Subjects rated their feelings of "Sluggish, Fatigued, Lazy" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 5.3 (4.2) | 12.9 (8.3)
  15 mg Cocaine | 13.4 (8.0) | 12.7 (6.7)
  45 mg Cocaine | 12.9 (6.8) | 7.7 (5.1)

22. Secondary Outcome: Peak Ratings of "Stimulated" on the Visual Analog Scale
Description: Subjects rated their feelings of "Stimulated" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 4.0 (3.1) | 4.2 (3.3)
  15 mg Cocaine | 18.7 (5.6) | 17.9 (5.7)
  45 mg Cocaine | 25.3 (7.6) | 32.3 (8.5)

23. Secondary Outcome: Peak Ratings of "Willing to Take Again" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Take Again" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.3 (2.4) | 3.2 (2.5)
  15 mg Cocaine | 27.7 (8.4) | 22.1 (8.3)
  45 mg Cocaine | 34.6 (11.0) | 43.4 (10.5)

24. Secondary Outcome: Peak Ratings of "Talkative, Friendly" on the Visual Analog Scale
Description: Subjects rated their feelings of "Talkative, Friendly" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: arbitary units on a Visual Analog Scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
arbitary units on a Visual Analog Scale
  0 mg Cocaine | 3.2 (2.6) | 2.0 (1.3)
  15 mg Cocaine | 11.7 (5.3) | 11.2 (4.8)
  45 mg Cocaine | 12.1 (4.6) | 21.8 (8.0)

25. Secondary Outcome: Peak Oral Temperature
Description: Oral temperature was measured with an automated monitor. Higher values represent greater temperature. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 3
Measure: Mean (Standard Error); unit: Degrees Fahrenheit
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
Degrees Fahrenheit
  0 mg Cocaine | 98.2 (0.1) | 98.3 (0.2)
  15 mg Cocaine | 98.3 (0.1) | 98.4 (0.2)
  45 mg Cocaine | 98.1 (0.1) | 98.4 (0.1)

26. Secondary Outcome: Peak Diastolic Blood Pressure
Description: Diastolic blood pressure was measured with an automated monitor. Higher values represent greater diastolic pressure. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 3
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
mmHg
  0 mg Cocaine | 74.3 (2.1) | 73.3 (3.1)
  15 mg Cocaine | 75.1 (2.5) | 74.6 (2.8)
  45 mg Cocaine | 77.6 (2.7) | 77.6 (2.4)

27. Secondary Outcome: Peak Heart Rate
Description: Heart rate was measured with an automated monitor. Higher values represent greater heart rate. Peak scores were calculated from multiple assessments for each cocaine dose under both buspirone and placebo conditions.
Time Frame: as for outcome 3
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 9 | 9
beats per minute
  0 mg Cocaine | 75.9 (3.6) | 79.7 (3.6)
  15 mg Cocaine | 79.9 (3.8) | 79.6 (4.6)
  45 mg Cocaine | 82.8 (2.7) | 89.3 (5.4)

ADVERSE EVENTS:
Groups:
- Buspirone: Subjects will be maintained on buspirone.
  Buspirone: Subjects will be maintained on oral buspirone (administered 3 times daily) or placebo for 6 days each during the study in random order. These subjects will be the same as those who are maintained on placebo (i.e., the study uses a within-subjects design).
- Placebo: Subjects will be maintained on placebo.
  Buspirone: Subjects will be maintained on oral buspirone (administered 3 times daily) or placebo for 6 days each during the study in random order.These subjects will be the same as those who are maintained on buspirone (i.e., the study uses a within-subjects design).
Arm/Group | Buspirone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No